CLINICAL TRIAL: NCT06781073
Title: An Multicenter, Randomized，Double-blind, Controlled Clinical Study of Nimotuzumab in Combined With First-line Chemotherapy for Treatment of IVB Stage,Rrecurrent or Persistent Cervical Squamous Cell Carcinoma
Brief Title: Nimotuzumab in Combined With Chemotherapy for Treatment of IVB Stage,Rrecurrent or Persistent Cervical Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPL-Nim-CC-2
Record Dates: First submitted 2023-07-24; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cervical Squamous Cell Carcinoma; Persistent
Keywords: Nimotuzumab; paclitaxel; cisplatin
MeSH Terms: interventions — nimotuzumab; Paclitaxel; Cisplatin; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab+TP(paclitaxel+cisplatin) (Experimental): experimental group
  Interventions: Drug: Nimotuzumab; Drug: Paclitaxel; Drug: Cisplatin
- Placebo + TP(paclitaxel+cisplatin) (Placebo Comparator): control group
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab in combined with chemotherapy period, 400mg, day1, administered intravenously before chemotherapy ,weekly, for 18 weeks; Maintenance period, 400mg, every two weeks until disease progression or intolerable toxicity , maximum duration is 60 weeks .
  Other Names: h-R3
  Arms: Nimotuzumab+TP(paclitaxel+cisplatin)
Drug: Paclitaxel — 175mg/m^2,for 3 hour,day1,21 days for a cycle ,until disease progression or toxicity，maximum duration is 6 cycles.
  Other Names: Paclitaxel Injection
Drug: Cisplatin — 50mg/m^2,day1orday2，21 days for a cycle ,until disease progression or toxicity,maximum duration is 6 cycles.
  Other Names: Cisplatin for Injection
Drug: Placebo — Placebo in combined with chemotherapy period, 400mg, day1, administered intravenously before chemotherapy ,weekly, for 18 weeks; Maintenance period, 400mg, every two weeks until disease progression or intolerable toxicity , maximum duration is 60 weeks .
  Other Names: Nimotuzumab Placebo
  Arms: Placebo + TP(paclitaxel+cisplatin)

SUMMARY:
This is an multicenter, randomized，double-blind, controlled clinical study. The purpose of the study is to evaluate the clinical efficacy and safety of Nimotuzumab combined with TP regimen (Paclitaxel + Cisplatin) for treatment of IVB stage, recurrent or persistent cervical squamous cell carcinoma .

DETAILED DESCRIPTION:
This clinical study is designed as an multicenter, randomized，double-blind, controlled clinical study to evaluate the clinical efficacy and safety of Nimotuzumab combined with TP regimen (Paclitaxel + Cisplatin) for treatment of IVB stage, recurrent or persistent cervical squamous cell carcinoma . The main endpoint is overall survival time, The secondary endpoint is no disease progression time,objective response rate and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and sign a consent form;
2. Age 18-75 years old ;
3. Histological diagnosis as cervical squamous cell carcinoma ;
4. Histologically and/or cytologically confirmed stage IVB or first recurrent or persistent cervical cancer (Mainly refers to the primary radiotherapy or concurrent chemoradiotherapy at least 3 months after the tumor remains or progress) and patients cannot receive surgery or radiation ;
5. Received taxoplatin + platinum combined chemotherapy stopped taking the drug for at least half a year, or received radiotherapy or concurrent chemoradiotherapy (cisplatin or cisplatin combined with 5-FU) for at least 3 months ;
6. According to the RECIST 1.1 criteria,there is at least one measurable lesion . The maximum diameter must meet the requirements : CT scan ≥10mm (CT scan thickness is less than 5mm); Clinical routine examination instrument 10mm (tumor lesions that cannot be accurately measured by diameter instruments should be recorded as unmeasurable), chest X-ray ≥20mm; Malignant lymph nodes: pathologically enlarged and measurable, single lymph node CT scan diameter ≥15mm (CT scan Layer thickness not more than 5mm) ;
7. Patients need to recover from toxic side effects (except decreased hemoglobin) of previous treatments (surgery, chemoradiotherapy, radiation therapy) to grade 1 or below （CTCAE 4.03）;
8. ECOG performance status 0-1 ;
9. Life expectancy of more than 3 months ;
10. Haemoglobin≥90g/L,white blood cell(WBC)≥4×109/L,Absolute neutrophil count≥1.5×109/L,platelet count≥100×109/L ;
11. TBIL≤1.5 ULN; ALK,AST and ALT≤2.5 ULN or ≤5 ULN(Liver metastasis) ; serum creatinine ≤ 1.5 ULN -

Exclusion Criteria:

1. Simple mediastinal or/and supraclavicular lymph node metastases ;
2. Bone metastases alone or multiple metastases with bone metastases requiring radiotherapy for pain relief ;
3. Patients with recurrence and metastasis after the end of the last administration of neoadjuvant chemotherapy or postoperative adjuvant chemotherapy < 6 months ;
4. Received anti-EGFR monoclonal antibody or small molecule TKI within 6 months prior to enrollment ;
5. Major surgery within 4 weeks or planned surgery or radiation therap ;
6. Participants in other interventional clinical trials within 1 month prior to informed consent ;
7. Neurological or psychiatric abnormalities that affect cognitive ability, including brain metastases ;
8. With clear peripheral neuropathy and related symptoms in the past;
9. Active clinical infection (>grade 2 NCI-CTCAE 4.03), active tuberculosis, and known or self-reported HIV infection or active hepatitis B or C ;
10. Severe respiratory system, blood system disease, intractable dysentery or intestinal cramps, intestinal obstruction, or poorly controlled diabetes ;
11. Uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg), congestive heart failure above NYHA Ⅲ, unstable angina or poorly controlled arrhythmia , circulatory diseases such as myocardial infarction before enrollment within 6 months ;
12. Have allergic reactions to study drugs and similar drugs ;
13. Pregnant or breast-feeding or refused to take contraceptive method;
14. Other malignant tumor;
15. Any other serious complications or dysfunction of the organ system, as judged by the investigator, will affect the safety of the patient or interfere with the evaluation of the test drug ; -

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 46 months
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 46 months
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD.
Objective Response Rate | Up to approximately 46 months
  This wil be evaluated by RECISIT 1.1 criteria.It is dependent on imaging evaluation which will be done every 6 weeks. ORR is the percent of the patient who is evaluated as complete response(CR) or partial response (PR),that is (CR+PR)%.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status Score | Baseline and up to approximately 46months
  The EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. The change from baseline in EORTC QLQ-C30 score will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) Score | Baseline and up to approximately 46months
  The EORTC QLQ-CX24 is a questionnaire that rates the symptoms common to women with cervical cancer and evaluates the impact of disease and/or treatments. The 24 items use a 4-point scale (1=not at all to 4=very much) and are classified into 3 multi-item scales, 11 items with symptom experience, 3 items with body image, and 4 items with sexual/ vaginal functioning. The other items of the questionnaire are lymphedema, peripheral neuropathy, menopausal symptom, sexual worry, sexual activity, and sexual enjoyment. The change from baseline in EORTC QLQ-CX24 score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: lingying wu, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital , Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No